CLINICAL TRIAL: NCT00390845
Title: A Double-blind Placebo-controlled Study of the Efficacy and Safety of the P38 Map Kinase Inhibitor SB681323 in Patients With Neuropathic Pain Following Nerve Trauma
Brief Title: P38 Mitogen-activated Protein (Map) Kinase Inhibitor (SB-681323)Study In Patients With Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: MKN106762
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pain, Neuropathic
Keywords: MAP kinase; SB681323; neuropathic pain; patients; P38; nerve trauma
MeSH Terms: conditions — Neuralgia | interventions — dilmapimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB681323 (Experimental): Patients with pain associated with peripheral nerve injury and/or compression will be recruited for this study.
  Interventions: Drug: SB681323
- Placebo (Experimental): Patients with pain associated with peripheral nerve injury and/or compression will be recruited for this study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB681323 — 15 milligrams (mg)/day
  Arms: SB681323
Drug: Placebo
  Arms: Placebo

SUMMARY:
This will be a double-blind, placebo controlled cross-over study. After enrolment and initial assessments, subjects will receive oral SB681323 or matching placebo for 14 days. SB681323 will be administered twice daily at a total daily dose of 7.5mg. Sufficient numbers of patients will be recruited to obtain 40 evaluable patients

ELIGIBILITY:
Inclusion criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:

Male or female subjects 18-80 years of age

* To be eligible, females patients must have a negative pregnancy test (i.e. serum beta hCG test) and be of:

  1. non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes any female who is post-menopausal. For the purposes of this study, post menopausal is defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. Postmenopausal status will be confirmed by serum FSH and oestradiol concentrations at screening. Surgical sterility will be defined as females who have had a hysterectomy and/or bilateral oophorectomy or tubal ligation.

OR b.childbearing potential and agree to commit to one of the protocol-approved methods of contraception, when used consistently and in accordance with both the product label and the instructions of a physician, as indicated below: i.oral contraceptive (combined or progestin only), and the same oral contraceptive regimen has been used for at least two months prior to study drug administration, and the same method continues throughout the study and through the follow-up phase of the study.

ii.progesterone implanted rods (Norplant ) inserted for at least two months prior to the study drug administration (but not beyond the third successive year following insertion) , and is continued throughout the study and through the follow-up phase of the study.

iii.an IUD, inserted by a qualified clinician, with published data showing that the highest expected failure rate is less than 1% per year (not all IUDs meet this criterion) Acceptable IUDs: TCu-380A (Paragard), TCU-380 Slimline (Gyne T Slimline), TCu-220C, MULTILOAD-250 (MLCu-250) and 375, NOVA T and CUNOVAT (Novagard), Levonorgesterol (LNG-20) Intra-uterine System (Mirena/Levonova), and FlexiGard 330/CuFix PP330 (Gynefix). The device must be inserted at least 2 weeks prior to the Screen visit, and remain throughout the study and through the follow-up phase of the study.

iv.injectable medroxyprogesterone acetate (e.g., Depo-Provera) and is on a stable dose for 2 months prior to Screen, throughout the study and through the follow-up phase of the study.

v.complete abstinence from intercourse from at least two weeks prior to Screen, throughout the treatment phase, and the follow-up phase.

vi.double barrier method if comprised of a spermicide with either a condom or diaphragm from at least two weeks prior to Screen, throughout the treatment phase, and the follow-up phase.

* A diagnosis of peripheral neuropathic pain:

  * focal neuropathic pain related to nerve injury caused by trauma or surgery not associated with ongoing infection (examples include post-thoracotomy syndrome, post-mastectomy syndrome, post-inguinal herniorrhaphy syndrome, post-radical neck dissection syndrome, traumatic mononeuropathies- bullet wounds, lacerations, road traffic accidents)
  * pain associated with lumbo-sacral radiculopathy; patients with radiculopathy will only be included if they have pain radiating below the knee and have loss of small fibre function as indicated by quantitative sensory testing (elevation of at least one sensory modality threshold in the symptomatic limb - warm sensation > 9.6 0C and cool sensation > 5.6 0C - in L4, L5 or S1 dermatomes) [Quraishi, 2004].
  * carpal tunnel syndrome (CTS); patients with CTS will only be included if there is evidence of loss of large and small fibre function (confirmed by an electrophysiological nerve conduction examination and by quantitative sensory testing - warm sensation > 5.2 0C and cool sensation > 4.5 0C - in median nerve territory (Anand et al., unpublished data).
  * location of pain consistent with the area innervated by the affected nerve(s), with or without other sensory symptoms in the affected area
  * at least three months duration
* Baseline pain intensity score averaging ≥ 4 during the three day prior to study start as reported on the 11 point pain intensity numerical rating scale. For CTS patients, peak daily pain will be ≥4 for at least 3 days prior to enrolment
* Subjects who have received nerve blocks or steroid injections for neuropathic pain may be included if their most recent nerve block was at least 4 weeks prior to randomisation.
* Body weight ≥ 50 kg (110 lbs) for men and ≥ 45 kg for women, Body Mass Index 18.5-35kg/m2.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within normal limits at screening.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Signed and dated written informed consent prior to admission to the study.

Exclusion criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Any clinically significant medical history or abnormality found on physical examination, laboratory assessment or ECG at screening which, in the opinion of the investigator, could interfere with the interpretation of efficacy or safety data or which otherwise would contraindicate participation in a clinical study, in particular:

  * subjects with non-neuropathic pain component involvement, mononeuropathy multiplex, or more than one cause or potential cause for pain symptoms (e.g. trigeminal neuralgia, painful diabetic neuropathy, central post-stroke pain, phantom limb pain, peripheral neuropathy due to alcoholism, malignancy, HIV, syphilis, drug abuse, vitamin deficiency, hypothyroidism, liver disease, toxic exposure, or chronic neck pain);
  * subjects with intractable pain of unknown origin or active infection in the area of nerve injury/compression;
  * subjects who have had extensive surgery in the treatment of their nerve injury;
  * history of Gilbert's syndrome or elevated bilirubin levels (total, direct or indirect) in a previous clinical study or at screening;
  * history of increased liver function tests (ALT, AST) above upper limit of normal in the past 6 months;
  * positive Hepatitis B surface antigen, positive Hepatitis C antibody or Hepatitis C nucleic acid result;
  * GI disorders that may interfere with safety assessments, e.g. diarrhoea.
* Recent start or change in dosing regimen (£1 month prior to screen) of any medication which, in the opinion of the Investigator, may interfere with pain assessments or introduce a risk of drug-drug interactions (e.g. glucocorticoids and some anticonvulsants, see Section 9.2, Prohibited Medications for details).
* Unable to refrain from excessive use medications (e.g. sedatives) that in the opinion of Investigator may interfere with efficacy or safety assessments (benzodiazepines prescribed as hypnotic sleep agents allowed). Subject is unable to discontinue topical analgesics prior to randomization and for the duration of the study. In the case of topical capsaicin this will be extended to 4 weeks.
* Subject is unable to refrain from nerve blocks during the study.
* Positive alcohol test or urine drug screen at screening.
* History of regular alcohol consumption exceeding an average weekly intake of > 21 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 14 units (or an average daily intake of greater than 2 units) for females.
* Consumption of grapefruit or grapefruit juice within seven days prior to the first dose of study medication.
* Donation of blood in excess of 500 mL within a 30-day period prior to dosing.
* Participation in a trial with any drug within 3 months before the start of the study or participation in a trial with a new chemical entity within 4 months before the start of the study.
* Pregnant or nursing female subjects.
* Known history of hypersensitivity or intolerance to paracetamol products.
* Inability or unwillingness to follow the instruction of the study protocol.
* Known hypersensitivity to capsaicin (if applicable)
* An unwillingness of male subjects to abstain from sexual intercourse with women; or unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception (as described in inclusion criterion for women) if the woman could become pregnant from the time of the first dose of investigational product until completion of the follow-up procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08-30 (Actual); Primary Completion 2008-08-11 (Actual); Study Completion 2008-08-11 (Actual)

PRIMARY OUTCOMES:
Mean average Daily Pain Intensity Numeric Rating Scale (PI-NRS) score over period | Day 1 to 14 of each treatment period
  Participants were asked to rate their overall pain intensity for the last 24 hours, daily before retiring to bed. This constituted the Daily Pain Score. The 11 point pain intensity numerical rating scale ranged from 0 to 10, where 0 represents "No pain" and 10 represents "Maximum pain imaginable". It was used for the subjective assessment of the pain. The score ranged from 0 to 10, where 0 represented absence of symptoms and higher score indicated more severe symptoms. The average daily pain over Week 1 (Day 7) was calculated as the mean of days 2 to 6 inclusive and for week 2 (Day 14), days 8 to 13 inclusive. Participants were instructed to record their daily pain score on a dairy card and calculations of average weekly pain scores were performed on the basis of diary cards review.

SECONDARY OUTCOMES:
Mean Current pain intensity (CPI) score using PI-NRS over period | Up to Day 14 of each treatment period
  The 11 point pain intensity numerical rating scale ranged from 0 to 10, where 0 represents "No pain" and 10 represents "Maximum pain imaginable". It was used for the subjective assessment of the pain. The score ranged from 0 to 10, where 0 represented absence of symptoms and higher score indicated more severe symptoms. Current pain was the pain intensity assessments that were carried out in the unit (at Day 7 and 14 of each treatment period), were recording of the pain intensity that the participant felt at the time.
Mean Quantitative Sensory Testing (QST) in cold pain, heat pain and warmth detection threshold on Day 14 | Day 14 of each treatment period
  A thermode was placed on skin of participant. Temperature of block was initially set to Baseline temperature of participant's skin (32 degree Celsius [°C]). For threshold measurement, temperature of thermode was gradually increased (for warm sensation and heat pain detection thresholds) or decreased (for cold sensation and cold pain thresholds) from Baseline (32°C) at rate of 1°C per second. Ramp was stopped and temperature of thermode was returned to Baseline by participant pushing a button on a response unit when threshold was reached. It was repeated 4 (sensation thresholds) or 3 times (pain thresholds) for each modality. Threshold temperatures and average values were recorded. If thermode temperature reached 50°C (heat pain) or 0°C (cold pain) without participant responding, ramp was stopped, temperature was returned to Baseline automatically to prevent skin injury. Respective cut-off temperature was then recorded for that trial. Recorded for affected and controlled area of skin.
Mean area of static touch allodynia | Day 1 of each treatment period
  Allodynia is defined as increased response of neurons on painful and repetitive, stimulation or pain in response when touched. Area of static allodynia was determined using a 26 g von Frey filament. In a non-painful area, investigator repeatedly applied filament perpendicularly to skin, exerting enough pressure to make filament bend slightly, each time closer to presumed border of allodynia. When participant reported sensation becoming more unpleasant or painful, point at which filament was contacting the painful area of skin was marked with a felt tip pen by investigator. At that point, if participant's painful area was on a limb, a total of four points (each 90° apart) were drawn in order to complete mapping. If participant's painful area was irregular, or on trunk or face, a total of 8 points (45° apart) was drawn in order to complete mapping. Area of static allodynia was calculated by transferring the points to an homunculus. Points were connected to form area of allodynia.
Mean area of dynamic touch allodynia | Day 1 of each treatment period
  Allodynia is defined as increased response of neurons on painful and repetitive, stimulation or pain in response to stroking lightly. Area of dynamic allodynia was determined using a one inch foam brush. In a non-painful area, investigator, exerted enough pressure to make foam brush bend slightly, would slowly move brush forward toward painful area of participant, at rate of 1 centimeter per second. When participant reported sensation becoming unpleasant or painful, point at which foam brush was contacting painful area of skin was marked with a felt tip pen by investigator. At that point, if participant's painful area was on a limb, a total of 4 points (each 90° apart) was drawn in order to complete mapping. If participant's painful area was irregular, or was in truncal or facial area, a total of 8 points (45° apart) were drawn in order to complete mapping. Area of dynamic allodynia was calculated by transferring points to an homunculus, were connected to form area of allodynia.
Mean intensity of static and dynamic touch allodynia | Day 1 of each treatment period
  Allodynia is defined as increased response of neurons on painful and repetitive, stimulation. Where static allodynia was pain in response when touched and dynamic allodynia was pain in response to stroking lightly. The intensity of static and dynamic allodynia was assessed using the 11 point numeric rating scale, where 0=no pain, 10=maximum pain imaginable. The score ranged from 0 to 10, where 0 represents absence of symptoms and higher score indicates more severe symptoms.
Number of participants with Global Impression of Change Scale scores over period | Up to Day 14 of each treatment period
  The Global Impression of Change scale was rated by the clinician and the participant for change in overall status as perceived by the clinician and as perceived by the participant, respectively. It was rated using a 7-point numerical rating scale where 1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse and 7=Very much worse. The scale ranged from 1 to 7, where 1 indicates best response and 7 indicates worst response. The assessments were done during the Visit to the unit on Day 7 and Day 14, 2 hours post-dose of each treatment period.
Number of participants who used rescue medication over period | Day 1 to 14 of each treatment period
  Any participant for whom the pain intensity became unacceptable during any stage of the study was permitted to initiate rescue analgesic therapy with the protocol defined rescue medication of paracetamol up to two 500 mg tablets BID (i.e., maximum paracetamol 2 g per 24 hour period). Total paracetamol use included rescue medication and also paracetamol consumed in over-the-counter remedies including cold, allergy, sleep and pain preparations. Participants were requested not to take any paracetamol up to 24 hours before a treatment Visit. The use of rescue medication was recorded on the diary cards by the participants and use of recue medication during the treatment visit was recorded in case report form (CRF). Data is reported for number of participants who used rescue medication.
Latency of contact heat-evoked potential stimulator (CHEPS) in the affected and control area | Day 1 of each treatment period
  Evoked potentials were planned to be recorded from midline electrodes. Responses from ten stimuli were planned to be recorded from each participant with the thermode placed over 3 sites -the lateral calf, lateral forearm and face (cheek). This involved a CHEPS with a thermode area of 572.5 mm^2 and a heating thermo foil covered with a 25 uncertainty of measurement (Um) layer of thermo conductive plastic. The thermode heating rate was planned at 70 °C per second and the cooling rate 40°C per second. The Baseline temperature was planned at 32 °C, destination temperature 51 °C, and stimulus interval was 7 seconds. Stimuli was planned to be applied to the dermatome of interest. The participant could withdraw at any time. The assessment was planned at the affected area and control area which was the mirror image site area. The assessment for this outcome measure was optional during the study and data was not collected for this outcome measure.
Amplitude of CHEPS in the affected and control area | Day 1 of each treatment period
  Evoked potentials were planned to be recorded from midline electrodes. Responses from ten stimuli was planned to be recorded from each participant with the thermode placed over 3 sites -the lateral calf, lateral forearm and face (cheek). This involved a CHEPS with a thermode area of 572.5 mm^2 and a heating thermo foil covered with a 25 uncertainty of measurement (Um) layer of thermo conductive plastic. The thermode heating rate was planned at 70 °C per second and the cooling rate 40°C per second. The Baseline temperature was planned at 32 °C, destination temperature 51 °C, and stimulus interval was 7 seconds. Stimuli was planned to be applied to the dermatome of interest. The participant could withdraw at any time. The assessment was planned at the affected area and control area which was the mirror image site area. The assessment for this outcome measure was optional during the study and data was not collected for this outcome measure.
Number of participants with skin biopsy results | 80 Days
  Assessemnt of capsaicin and heat receptor TRPV1 immunoreactivity and mechanism-related markers (NGF, CGRP) in skin biopsies was optional outcome measure, planned to be conducted on participants proceeding to surgery. However the data for this outcome measure was not collected and result summary was not produced.
Number of participants with any adverse event (AE), serious adverse event (SAE) or death | Up to Follow-up (80 Days)
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of participants with clinical chemistry values of potential clinical concern (PCC) during treatment period | Day 1 to Day 14 of each treatment period
  The parameters of clinical chemistry included sodium, potassium, urea, creatinine, total protein, albumin, total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), gamma glutamyl transferase (GGT), lactate dehydrogenase (LDH), calcium, magnesium, phosphate, cholesterol, high density lipoprotein (HDL) cholesterol, triglycerides, glucose and creatinine kinase. The assessments were done at Day 1, 7 and 14 of each treatment period. Only those parameters for which at least one value of PCC was reported are summarized
Number of participants with hematology values of PCC during treatment period | Day 1 to Day 14 of each treatment period
  The parameters of hematology included hemoglobin (Hb), packed cell volume (PCV), mean cell hemoglobin (MCH), mean cell hemoglobin concentration (MCHC), red blood cell count (RBC), white blood cell count (WBC), platelets, differential WBC count and examination of film. The assessments were done at Day 1, 7 and 14 of each treatment period. Only those parameters for which at least one value of PCC was reported are summarized.
Number of participants with vital sign values of PCC during treatment period | Day 1 to Day 14 of each treatment period
  Vital signs assessment included heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP), done while participant lying supine and having rested in this position for at least 10 minutes before each reading. Criteria for vital sign values meeting PCC included: SBP < 85 and > 160 millimeters of mercury (mmHg) and increase or decrease from Baseline >= 20 and >= 40 mmHg; DBP < 45 and > 100 mmHg and increase or decrease from Baseline >= 10 and >= 20 mmHg; HR < 40 and > 110 beats per minute (bpm) and increase or decrease from Baseline >= 15 and >= 30 bpm. The assessments were done at Day 1, Day 7 and Day 14 (pre dose and 1.5 hour post dose) of each treatment period. Only those parameters for which at least one value of PCC was reported are summarized.
Number of participants with normal and abnormal (not clinically significant [NCS] and clinically significant [CS]) electrocardiogram (ECG) findings | Day 1 to Day 14 of each treatment period
  Full 12 lead ECGs were recorded using an ECG machine that automatically calculated the HR and measured PR, QRS, QT, Bazzette formula corrected QT (QTcb) interval and Fridericia formula corrected QT (QTcF) interval. Overall ECG findings were summarized at Day 1, Day 7 and Day 14 of each treatment period (pre-dose and 1.5 hour post-dose). Normal and abnormal ECG findings were categorized. The abnormal PCC ranges were: absolute QTc interval >450 msec and increase from baseline QTc >=60 and <=59; PR interval <110 and >220 msec; QRS interval <75 and >110 msec.
Number of pregnancies in females of child bearing potential during treatment period | Up to Follow-up (80 days)
  Urine human chorionic gonadotrophin (β-hCG) pregnancy test was performed in all female participants of childbearing potential only at Day 1 and Day 14 of each treatment period and Follow-up. In the case of a positive urine β-hCG test, pregnancy was confirmed with a serum β-hCG test.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Australia (2):
  - GSK Investigational Site, Broadmeadow, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
- Germany (4):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
- GSK Investigational Site, Moscow, Russia
- United Kingdom (5):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Solihull, West Midlands
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London